CLINICAL TRIAL: NCT03981042
Title: Comparison Between the Neuromuscular Blockade Onset Monitoring and the Expectation of a Fixed Delay After Curarization on the Quality of Laryngoscopy During Intubation in Elective Surgery (MONITURARE)
Acronym: MONITURARE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2019-A00667-50
Record Dates: First submitted 2019-04-24; First posted 2019-06-10 (Actual); Last update posted 2019-10-21 (Actual); Status verified 2019-10

CONDITIONS: Laryngoscopy; Anesthesic Aduction; Neuromuscular Blockade; Monitoring
Keywords: laryngoscopy; anesthesic aduction; neuromuscular blockade monitoring

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): waiting for a 3-minute delay after injection of the atracurium before laryngoscopy
- Monitoring group (Experimental): waiting for the TOF ratio at 0 at the corrugator supercilli before laryngoscopy
  Interventions: Device: Monitoring

INTERVENTIONS:
Device: Monitoring — After the anesthetic induction with sufentanil, propofol and atracurium, patients will be ventilated with mask until:
  - Monitoring group: TOF ratio at the corrugator supercilli will be measured every 15 s after injection of atracurium. When TOF ratio reach 0, laryngoscopy with intubation will be performed
  Arms: Monitoring group

SUMMARY:
During anesthetic induction, the relevance of neuromuscular blockade (NMB) onset monitoring cannot be asserted and its superiority over waiting for a fixed delay (corresponding to pharmacokinetic knowledge of the neuromuscular blocking agent used) has not been proven. However, many studies have shown a large inter-individual variability on the delay of the NMB onset. The main objective of othe investigator's study is to compare the quality of laryngoscopy during intubation between the NMB onset monitoring and the expectation of a fixed delay after curarization

DETAILED DESCRIPTION:
French guidelines on curarization, updated in 2018, do not recommend the NMB onset monitoring due to a lack of data in the literature. Thus, the interest of monitoring cannot be asserted and its superiority over waiting for a fixed delay has not been proven.

Due to a large inter-individual variability on the delay of the NMB onset after administration of atracurium, the relevance of monitoring NMB during an anesthetic induction should be assessed to improve the quality of laryngoscopy.

In case of monitoring, the experts recommend monitoring the NMB onset at the corrugator supercilli because it reflects neuromuscular blockade at the laryngeal adductor muscles.

During the pre-anaesthetic visit, patients will be enrolled after inform consent.

Patients will be randomized in two groups, control group (waiting for a 3-minute delay after injection of atracurium) or monitoring group (waiting for the TOF ratio at 0 at the corrugator supercilli).

Anesthetic induction will be performed with sufentanil, propofol and atracurium. After laryngoscopy, the primary outcome will be evaluated using Copenhagen score.

Patients will be followed up until they leave the recovery room..

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥ 18 years), both sexes
* Any elective surgery requiring injection of atracurium
* Free patient, without guardianship or subordination
* Patients with a social security coverage
* Informed and signed consent after clear and fair information

Exclusion Criteria:

* Rapid sequence induction
* Predictable difficult intubation
* Use of a neuromuscular blockade agent other than atracurium
* Known contraindication to a neuromuscular blockade agent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2019-06-14 (Actual); Primary Completion 2019-08-02 (Actual); Study Completion 2019-08-02 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is the assessment of the Copenhagen score modified collected during the anesthetic induction after the intubation. | Few minutes after intubation (about 5 minutes)
  The primary endpoint is the assessment of the Copenhagen score modified collected during the anesthetic induction after the intubation.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU, Poitiers, France